CLINICAL TRIAL: NCT06252558
Title: Do Symbiotics Provide Helpful Benefits in Gastrointestinal Related Issues in Weight Loss Surgery Patients?
Brief Title: Symbiotic Use in Post-Bariatric Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Florida (Other)
Collaborators: Celebrate Nutritional Supplements (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2089663-1
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric surgery; symbiotic; prebiotics; probiotics; weight loss surgery
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symbiotic Group (Experimental): An over-the counter, once daily symbiotic capsule including: 15 billion CFU probiotic blend and 250mg of prebiotic.
  Interventions: Dietary Supplement: Symbiotic
- Fiber Group (Placebo Comparator): Once daily capsule of microcrystalline cellulose.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Symbiotic — One-a-day administration of a capsule supplement containing:15 billion CFU probiotic blend (Lactobacillus acidophilus La-14, Bifidobacterium longum BB536, Lactobacillus acidophilus NCFM, Lactobacillus rhamnosus GG, Lactobacillus gasseri Lg-36) and 250mg of chicory root inulin.
  Other Names: Celebrate Balance Probiotic Plus Prebiotic
  Arms: Symbiotic Group
Dietary Supplement: Placebo — Daily fiber capsule containing microcrystalline cellulose
  Arms: Fiber Group

SUMMARY:
The purpose of this double blind, randomized control trial would be to test the efficacy of a once daily, multi strain symbiotic on gut health changes in weight loss surgery patients by testing stool samples prior to administration and then three months post administration of the symbiotic to monitor any changes in bacteria in the stool samples. Study participants will also complete a survey that evaluates their bowel habits, stool consistency, and gastrointestinal related symptoms.

DETAILED DESCRIPTION:
The topic of interest is the gut microbiome and the impact of symbiotics (prebiotics coupled with probiotics) on gut health after weight loss surgeries due to surgical alterations of the stomach and bowels as a result of the procedures. Symbiotics provide positive gut health benefits, ie. improvement in bowel function and reduction in gastrointestinal distress symptoms such as bloating. However, when conducting a literature review on probiotics/prebiotics, most of the research studies have poor quality and do not cite the quantity of each strain being studied. To date, no research has been conducted on symbiotic administration in post bariatric surgery patients and their relationship regarding improvements in gastrointestinal symptoms.

There is no standard dose recommended for probiotics. Each strain should be given at a dose that has shown to be effective at providing a health benefit to the host through clinical trials. However, no clear criteria has been established to determine what classifies as effective and what health benefits are considered clinically relevant. Most healthcare organizations recommend between 1 to 20 x 109 colony forming units (CFU)/ day for adults. In many cases, higher dosages have been shown to be more effective, but a clear dose-dependent response has not been identified and a "more is better" philosophy does not apply to all strains. Therefore, one rule states that "If a product contains multiple strains, then each strain should be present at levels of 109 to ensure effectiveness."

The primary objective of this study would be to determine the efficacy of symbiotic administration for improving gastrointestinal health in weight loss surgery patients. This study would test the efficacy of a once daily, multi strain symbiotic on gut health changes in weight loss surgery patients, twelve months or greater post-surgery, by testing stool samples prior to administration and then three months after administration of the symbiotic to monitor any changes in bacteria in the stool samples. Study participants will also complete a survey that evaluates their bowel habits, stool consistency, and gastrointestinal symptoms prior and post symbiotic administration.

ELIGIBILITY:
Inclusion Criteria:

* 12 months or greater post malabsorptive weight loss procedure

Exclusion Criteria:

* LapBand or Intra-gastric balloon patients due to lack of surgical alteration to gut
* Individuals who have not had an approved weight loss procedure
* Individuals with impaired gastrointestinal function which would impair ingestion of oral supplement
* Individuals with impaired gastrointestinal function which would impair ability to collect stool sample
* Inability to comprehend and complete assessment tools
* Inability to adhere to 90-day capsule supplement administration
* Currently taking daily probiotic, prebiotic, or symbiotic supplement
* Currently taking antibiotic treatment from physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symbiotic Changes in Stool Samples | 90 days
  The primary objective will be to test the efficacy of a once daily, multi-strain symbiotic on gut health changes in weight loss surgery patients by testing stool samples prior to administration and then three months after administration of a symbiotic or placebo. Chi-square tests will be performed to show associations between symbiotic intake and stool bacteria diversity and concentrations.

SECONDARY OUTCOMES:
Bristol Stool Scale Weekly Changes | 12 weeks
  Participants will complete a weekly Bristol Stool Scale that identifies their overall stool consistency for the week.Participants will complete this tool weekly and SPSS software will be used to conduct an independent t-test of mean changes to evaluate the difference in stool form. Total scores can range from 7 through 49, with scores closest to 24.5 representing normal stool form. The comparisons of these tests will be able to provide statistical relevance on the usage of symbiotic supplementation in normal stool form.
Frequency of Weekly Stools | 12 weeks
  Participants will complete a weekly survey that identifies the amount of stools produced the week prior. Independent t-test will be performed to show changes in stool frequency.
Gastrointestinal Related Symptoms | 12 weeks
  A final Chi-square test of association will be performed using SPSS software to test whether there is a relationship between symbiotic intake and reduction in GI related symptoms. P-values of 0.05 or lower will be used to prove statistical significance for all tests performed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lim Y, Boster J. Obesity and Comorbid Conditions. StatPearls. Published online October 25, 2021. Accessed March 28, 2022. https://www.ncbi.nlm.nih.gov/books/NBK574535/
- [Background] Obesity Medicine Association. AMA Classifies Obesity as a Disease | Obesity Medicine AssociationMain. Published June 19, 2013. Accessed May 2, 2022.
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Ward ZJ, Bleich SN, Cradock AL, Barrett JL, Giles CM, Flax C, Long MW, Gortmaker SL. Projected U.S. State-Level Prevalence of Adult Obesity and Severe Obesity. N Engl J Med. 2019 Dec 19;381(25):2440-2450. doi: 10.1056/NEJMsa1909301. PMID 31851800
- [Background] Bhutani S, vanDellen MR, Cooper JA. Longitudinal Weight Gain and Related Risk Behaviors during the COVID-19 Pandemic in Adults in the US. Nutrients. 2021 Feb 19;13(2):671. doi: 10.3390/nu13020671. PMID 33669622
- [Background] Kim J, Eisenberg D, Azagury D, Rogers A, Campos GM. American Society for Metabolic and Bariatric Surgery position statement on long-term survival benefit after metabolic and bariatric surgery. Surg Obes Relat Dis. 2016 Mar-Apr;12(3):453-459. doi: 10.1016/j.soard.2015.11.021. Epub 2015 Nov 27. PMID 26944548
- [Background] American Society of Metabolic and Bariatric Surgery. Access to Care Fact Sheet. Published 2011. Accessed March 29, 2022. https://asmbs.org/resources/access-to-care-fact-sheet
- [Background] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, De Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society for Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO): Indications for Metabolic and Bariatric Surgery. Surg Obes Relat Dis. 2022 Dec;18(12):1345-1356. doi: 10.1016/j.soard.2022.08.013. Epub 2022 Oct 21. PMID 36280539
- [Background] Carter J, Chang J, Birriel TJ, Moustarah F, Sogg S, Goodpaster K, Benson-Davies S, Chapmon K, Eisenberg D. ASMBS position statement on preoperative patient optimization before metabolic and bariatric surgery. Surg Obes Relat Dis. 2021 Dec;17(12):1956-1976. doi: 10.1016/j.soard.2021.08.024. Epub 2021 Sep 3. No abstract available. PMID 34629296
- [Background] Youdim A. Bariatric Surgery. Merck Manual Professional Version. Published August 2021. Accessed April 17, 2022. https://www.merckmanuals.com/professional/nutritional-disorders/obesity-and-the-metabolic-syndrome/bariatric-surgery
- [Background] Stefater MA, Wilson-Perez HE, Chambers AP, Sandoval DA, Seeley RJ. All bariatric surgeries are not created equal: insights from mechanistic comparisons. Endocr Rev. 2012 Aug;33(4):595-622. doi: 10.1210/er.2011-1044. Epub 2012 May 1. PMID 22550271
- [Background] Center for Disease Control and Prevention. Adult Obesity Facts. Published September 30, 2021. Accessed March 28, 2022. https://www.cdc.gov/obesity/data/adult.html
- [Background] Owens DK. Interpretation of cost-effectiveness analyses. J Gen Intern Med. 1998 Oct;13(10):716-7. doi: 10.1046/j.1525-1497.1998.00211.x. No abstract available. PMID 9798822
- [Background] Weight Management Dietetic Practice Group. Pocket Guide to Bariatric Surgery. Third Edition. (Isom KA, Majumdar MC, eds.).; 2022.
- [Background] International Federation of Surgery for Obesity. Gastric Bypass Surgery. Accessed April 12, 2022. https://www.ifso.com/roux-en-y-gastric-bypass/
- [Background] International Federation of Surgery for Obesity. Biliopancreatic Diversion. Accessed April 12, 2022. https://www.ifso.com/bilio-pancreatic-diversion-with-duodenal-switch/
- [Background] International Federation of Surgery for Obesity. Laparoscopic Single Anastomosis Duodenal-Ileal bypass with Sleeve (SADI-S). Accessed April 12, 2022. https://www.ifso.com/single-anastomosis-duodenal-Ileal-bypass-with-sleeve/
- [Background] Arterburn DE, Telem DA, Kushner RF, Courcoulas AP. Benefits and Risks of Bariatric Surgery in Adults: A Review. JAMA. 2020 Sep 1;324(9):879-887. doi: 10.1001/jama.2020.12567. PMID 32870301
- [Background] American Society for Metabolic and Bariatric Surgery. Estimate of Bariatric Surgery Numbers, 2011-2019. Published March 2021. Accessed April 11, 2022.
- [Background] Mechanick JI, Apovian C, Brethauer S, Garvey WT, Joffe AM, Kim J, Kushner RF, Lindquist R, Pessah-Pollack R, Seger J, Urman RD, Adams S, Cleek JB, Correa R, Figaro MK, Flanders K, Grams J, Hurley DL, Kothari S, Seger MV, Still CD. CLINICAL PRACTICE GUIDELINES FOR THE PERIOPERATIVE NUTRITION, METABOLIC, AND NONSURGICAL SUPPORT OF PATIENTS UNDERGOING BARIATRIC PROCEDURES - 2019 UPDATE: COSPONSORED BY AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS/AMERICAN COLLEGE OF ENDOCRINOLOGY, THE OBESITY SOCIETY, AMERICAN SOCIETY FOR METABOLIC & BARIATRIC SURGERY, OBESITY MEDICINE ASSOCIATION, AND AMERICAN SOCIETY OF ANESTHESIOLOGISTS - EXECUTIVE SUMMARY. Endocr Pract. 2019 Dec;25(12):1346-1359. doi: 10.4158/GL-2019-0406. Epub 2019 Nov 4. PMID 31682518
- [Background] Tabesh MR, Maleklou F, Ejtehadi F, Alizadeh Z. Nutrition, Physical Activity, and Prescription of Supplements in Pre- and Post-bariatric Surgery Patients: a Practical Guideline. Obes Surg. 2019 Oct;29(10):3385-3400. doi: 10.1007/s11695-019-04112-y. PMID 31367987
- [Background] Lysen LK, Isreal DA. Nutrition in Weight Management. In: Mahan KL, Escott-Stump S, Raymond JL, eds. Krause's Food and Nutrition Care Process. 13th ed. Elsevier; 2012:462-488.
- [Background] Sherf Dagan S, Goldenshluger A, Globus I, Schweiger C, Kessler Y, Kowen Sandbank G, Ben-Porat T, Sinai T. Nutritional Recommendations for Adult Bariatric Surgery Patients: Clinical Practice. Adv Nutr. 2017 Mar 15;8(2):382-394. doi: 10.3945/an.116.014258. Print 2017 Mar. PMID 28298280
- [Background] Sawaya RA, Jaffe J, Friedenberg L, Friedenberg FK. Vitamin, mineral, and drug absorption following bariatric surgery. Curr Drug Metab. 2012 Nov;13(9):1345-55. doi: 10.2174/138920012803341339. PMID 22746302
- [Background] Sherf-Dagan S, Buch A, Ben-Porat T, Sakran N, Sinai T. Vitamin E status among bariatric surgery patients: a systematic review. Surg Obes Relat Dis. 2021 Apr;17(4):816-830. doi: 10.1016/j.soard.2020.10.029. Epub 2020 Nov 10. PMID 33323330
- [Background] World Gastroenterology Organisation (WGO). WGO Practice Guidelines Probiotics and Prebiotics. February 2017. https://www.worldgastroenterology.org/guidelines/probiotics-and-prebiotics
- [Background] International Scientific Association for Probiotics and Prebiotics. The ISAPP quick guide to probiotics for health professionals: History, efficacy, and safety. December, 2019. https://isappscience.org/for-clinicians/resources/probiotics/#toggle-id-1
- [Background] Sweeney TE, Morton JM. The human gut microbiome: a review of the effect of obesity and surgically induced weight loss. JAMA Surg. 2013 Jun;148(6):563-9. doi: 10.1001/jamasurg.2013.5. PMID 23571517
- [Background] Zhang Y, Yan T, Xu C, Yang H, Zhang T, Liu Y. Probiotics Can Further Reduce Waist Circumference in Adults with Morbid Obesity after Bariatric Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2021 Apr 1;2021:5542626. doi: 10.1155/2021/5542626. eCollection 2021. PMID 33859706
- [Background] Wang Y, Wu XT, Chen J. Effect of Probiotic Supplementation on Weight Loss, Inflammatory Factors, and Metabolic Effects in Patients Undergoing Bariatric Surgery. Obes Surg. 2022 May;32(5):1779-1782. doi: 10.1007/s11695-022-05974-5. Epub 2022 Mar 4. No abstract available. PMID 35243603
- [Background] Seganfredo FB, Blume CA, Moehlecke M, Giongo A, Casagrande DS, Spolidoro JVN, Padoin AV, Schaan BD, Mottin CC. Weight-loss interventions and gut microbiota changes in overweight and obese patients: a systematic review. Obes Rev. 2017 Aug;18(8):832-851. doi: 10.1111/obr.12541. Epub 2017 May 19. PMID 28524627
- [Background] Farup PG, Valeur J. Changes in Faecal Short-Chain Fatty Acids after Weight-Loss Interventions in Subjects with Morbid Obesity. Nutrients. 2020 Mar 18;12(3):802. doi: 10.3390/nu12030802. PMID 32197409
- [Background] Zhang H, DiBaise JK, Zuccolo A, Kudrna D, Braidotti M, Yu Y, Parameswaran P, Crowell MD, Wing R, Rittmann BE, Krajmalnik-Brown R. Human gut microbiota in obesity and after gastric bypass. Proc Natl Acad Sci U S A. 2009 Feb 17;106(7):2365-70. doi: 10.1073/pnas.0812600106. Epub 2009 Jan 21. PMID 19164560
- [Background] Fouladi F, Brooks AE, Fodor AA, Carroll IM, Bulik-Sullivan EC, Tsilimigras MCB, Sioda M, Steffen KJ. The Role of the Gut Microbiota in Sustained Weight Loss Following Roux-en-Y Gastric Bypass Surgery. Obes Surg. 2019 Apr;29(4):1259-1267. doi: 10.1007/s11695-018-03653-y. PMID 30604078
- [Background] Zuo HJ, Xie ZM, Zhang WW, Li YR, Wang W, Ding XB, Pei XF. Gut bacteria alteration in obese people and its relationship with gene polymorphism. World J Gastroenterol. 2011 Feb 28;17(8):1076-81. doi: 10.3748/wjg.v17.i8.1076. PMID 21448362
- [Background] Woodard GA, Encarnacion B, Downey JR, Peraza J, Chong K, Hernandez-Boussard T, Morton JM. Probiotics improve outcomes after Roux-en-Y gastric bypass surgery: a prospective randomized trial. J Gastrointest Surg. 2009 Jul;13(7):1198-204. doi: 10.1007/s11605-009-0891-x. Epub 2009 Apr 18. PMID 19381735
- [Background] Aron-Wisnewsky J, Prifti E, Belda E, Ichou F, Kayser BD, Dao MC, Verger EO, Hedjazi L, Bouillot JL, Chevallier JM, Pons N, Le Chatelier E, Levenez F, Ehrlich SD, Dore J, Zucker JD, Clement K. Major microbiota dysbiosis in severe obesity: fate after bariatric surgery. Gut. 2019 Jan;68(1):70-82. doi: 10.1136/gutjnl-2018-316103. Epub 2018 Jun 13. PMID 29899081
- [Background] Calikoglu F, Barbaros U, Uzum AK, Tutuncu Y, Satman I. The Metabolic Effects of Pre-probiotic Supplementation After Roux-en-Y Gastric Bypass (RYGB) Surgery: a Prospective, Randomized Controlled Study. Obes Surg. 2021 Jan;31(1):215-223. doi: 10.1007/s11695-020-04894-6. Epub 2020 Aug 15. PMID 32803709
- [Background] Kazzi F, Daher N, Zimmerman G, Garcia M, Schmidt N, Scharf K. Effect of Bacillius Coagulans and Galactomannans on Obese Patients Undergoing Sleeve Gastrectomy, A Randomized-Controlled Clinical Trial. Altern Ther Health Med. 2021 Jun;27(S1):138-145. PMID 29874199
- [Background] Shoaib M, Shehzad A, Omar M, Rakha A, Raza H, Sharif HR, Shakeel A, Ansari A, Niazi S. Inulin: Properties, health benefits and food applications. Carbohydr Polym. 2016 Aug 20;147:444-454. doi: 10.1016/j.carbpol.2016.04.020. Epub 2016 Apr 8. PMID 27178951
- [Background] Anderson JW, Baird P, Davis RH Jr, Ferreri S, Knudtson M, Koraym A, Waters V, Williams CL. Health benefits of dietary fiber. Nutr Rev. 2009 Apr;67(4):188-205. doi: 10.1111/j.1753-4887.2009.00189.x. PMID 19335713
- [Background] Sinn DH, Song JH, Kim HJ, Lee JH, Son HJ, Chang DK, Kim YH, Kim JJ, Rhee JC, Rhee PL. Therapeutic effect of Lactobacillus acidophilus-SDC 2012, 2013 in patients with irritable bowel syndrome. Dig Dis Sci. 2008 Oct;53(10):2714-8. doi: 10.1007/s10620-007-0196-4. Epub 2008 Feb 15. PMID 18274900
- [Background] Maria Remes Troche J, Coss Adame E, Angel Valdovinos Diaz M, Gomez Escudero O, Eugenia Icaza Chavez M, Antonio Chavez-Barrera J, Zarate Mondragon F, Antonio Ruiz Velarde Velasco J, Rafael Aceves Tavares G, Antonio Lira Pedrin M, Cerda Contreras E, Carmona Sanchez RI, Guerra Lopez H, Solana Ortiz R. Lactobacillus acidophilus LB: a useful pharmabiotic for the treatment of digestive disorders. Therap Adv Gastroenterol. 2020 Nov 24;13:1756284820971201. doi: 10.1177/1756284820971201. eCollection 2020. PMID 33281937
- [Background] Kailasapathy K, Chin J. Survival and therapeutic potential of probiotic organisms with reference to Lactobacillus acidophilus and Bifidobacterium spp. Immunol Cell Biol. 2000 Feb;78(1):80-8. doi: 10.1046/j.1440-1711.2000.00886.x. PMID 10651933
- [Background] Preston K, Krumian R, Hattner J, de Montigny D, Stewart M, Gaddam S. Lactobacillus acidophilus CL1285, Lactobacillus casei LBC80R and Lactobacillus rhamnosus CLR2 improve quality-of-life and IBS symptoms: a double-blind, randomised, placebo-controlled study. Benef Microbes. 2018 Sep 18;9(5):697-706. doi: 10.3920/BM2017.0105. Epub 2018 Jun 11. PMID 29888656
- [Background] Picard C, Fioramonti J, Francois A, Robinson T, Neant F, Matuchansky C. Review article: bifidobacteria as probiotic agents -- physiological effects and clinical benefits. Aliment Pharmacol Ther. 2005 Sep 15;22(6):495-512. doi: 10.1111/j.1365-2036.2005.02615.x. PMID 16167966
- [Background] Bouvier M, Meance S, Bouley C, Berta JL, Grimaud JC. Effects of consumption of a milk fermented by the probiotic strain Bifidobacterium animalis DN-173 010 on colonic transit times in healthy humans. Bioscience Microflora 2001; 20: 43-48.
- [Background] Ringel-Kulka T, McRorie J, Ringel Y. Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate the Benefit of the Probiotic Bifidobacterium infantis 35624 in Non-Patients With Symptoms of Abdominal Discomfort and Bloating. Am J Gastroenterol. 2017 Jan;112(1):145-151. doi: 10.1038/ajg.2016.511. Epub 2016 Nov 15. PMID 27845337
- [Background] Kligler B, Cohrssen A. Probiotics. Am Fam Physician. 2008 Nov 1;78(9):1073-8. PMID 19007054
- [Background] Probiotics: Fact Sheet for Health Professionals. National Institute of Health Office of Dietary Supplements.
- [Background] Ouwehand AC. A review of dose-responses of probiotics in human studies. Benef Microbes. 2017 Apr 26;8(2):143-151. doi: 10.3920/BM2016.0140. Epub 2016 Dec 23. PMID 28008787